CLINICAL TRIAL: NCT03562949
Title: A Randomized, Multiple-Dose, Placebo-Controlled, Multi-Center Study Comparing Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg to QVAR® 40 mcg (Beclomethasone Dipropionate HFA), Inhalation Aerosol in Treatment of Subjects With Asthma
Brief Title: A BE Study to Compare Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg and QVAR® 40 mcg, Inhalation Aerosol
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient investigational product
Sponsor: Amneal Ireland Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI-BDP-001
Record Dates: First submitted 2018-05-25; First posted 2018-06-20 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Test Product (Experimental): Test Product, 40 mcg, 2 x daily
  Interventions: Drug: Test Product
- Reference Product (Active Comparator): Reference Product, 40 mcg, 2 x daily
  Interventions: Drug: Reference Product
- Placebo (Placebo Comparator): Placebo Product 2 x daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Test Product — Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg
  Arms: Test Product
Drug: Reference Product — QVAR® 40 mcg (Beclomethasone Dipropionate HFA)
  Other Names: QVAR
  Arms: Reference Product
Drug: Placebo — Placebo Product
  Arms: Placebo

SUMMARY:
To compare the efficacy and safety profiles of Beclomethasone dipropionate Inhalation Aerosol, 40 mcg (test product) and QVAR 40 mcg (beclomethasone dipropionate HFA), Inhalation Aerosol (reference product) and to demonstrate that the efficacy of the 2 active products is superior to that of placebo in the treatment of subjects with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female subjects of non-childbearing or of childbearing potential committing to consistent and correct use of an acceptable method of birth control.
* Diagnosis of asthma as defined by the National Asthma Education and Prevention Program at least 12 months prior to screening.
* Pre-bronchodilator FEV1 of >45% and <85% of predicted value during the screening visit and on the first day of treatment.
* >15% and >0.20 L reversibility of FEV1 within 30 minutes following 360 mcg of albuterol inhalation (pMDI).
* Patients should be stable on their chronic asthma treatment regimen for at least four weeks prior to enrollment.
* Currently non-smoking; had not used tobacco products (i.e., cigarettes, cigars, pipe tobacco) within the past year, and having had <10 pack-years of historical use.
* Ability to replace current short-acting β agonist (SABAs) with salbutamol/albuterol inhaler for use as needed for the duration of the study. Subjects should be able to withhold all inhaled SABAs for at least six hours prior to lung function assessments on study visits.
* Ability to discontinue their asthma medications (inhaled corticosteroids and long-acting β agonists) during the run-in period and for remainder of the study.
* Willingness to give their written informed consent to participate in the study.

Exclusion Criteria:

* Life-threatening asthma, defined as a history of asthma episodes(s) requiring intubation, and/or associated with hypercapnia, respiratory arrest or hypoxic seizures, asthma related syncopal episode(s), or hospitalizations within the past year prior to the screening or during the run-in period.
* Significant respiratory disease other than asthma (COPD, interstitial lung disease, etc.)
* Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that, in the opinion of the investigator, would put the patient at risk through study participation, or would affect the study analyses if the disease exacerbates during the study.
* Viral or bacterial, upper or lower respiratory tract infection, or sinus, or middle ear infection within four weeks prior to the screening, during the run-in period, or on the day of treatment.
* Hypersensitivity to any sympathomimetic drug (e.g., albuterol) or any inhaled, intranasal, or systemic corticosteroid therapy.
* Patients receiving β2-blockers, anti-arrhythmics, anti-depressants, and monoamine oxidase inhibitors within 4 weeks prior to the screening.
* Patients who required systemic corticosteroids (for any reason) within the past 2 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted, pre-dose FEV1 on the last day of the 4-week treatment period | 4 weeks
  FEV1 measured in the morning prior dosing of inhaled medications on the last day of the 4-week treatment. The primary endpoint should be baseline adjusted (change from baseline).

OTHER OUTCOMES:
Number and type of adverse events | Minimum of a 2-week run-in period followed by a 4-week treatment period
  To investigate the safety and tolerability of Beclomethasone Dipropionate Inhalation Aerosol, 40 mcg and QVAR® 40 mcg, Inhalation Aerosol in the target population.

CONTACTS AND LOCATIONS:
Overall Officials: Irshad Haque, Study Director — Amneal Pharmaceuticals, LLC
Locations (12):
- United States (12):
  - Beach Clinical Research, Inc., Huntington Beach, California
  - Downtown La Research Center, Los Angeles, California
  - Moonshine Research Center, Doral, Florida
  - Hope Clinical Trials, Inc., Miami, Florida
  - San Marcus Research Clinic, Inc., Miami Lakes, Florida
  - Advanced Research for Health Improvement, Naples, Florida
  - Florida Institute for Clinical Research, Orlando, Florida
  - Innovation Research Center, Palmetto Bay, Florida
  - Florida Premier Research Institute, Winter Park, Florida
  - Monroe BioMedical Research, Monroe, North Carolina
  - TTS Research, Boerne, Texas
  - PCP for Life/ Mercury Clinical Research, Splendora, Texas